CLINICAL TRIAL: NCT03419143
Title: Abatacept - Long-Term Real-Life Experience in Psoriatic Arthritis (PsA) in Germany: an Observational Study (ALTEA)
Brief Title: Safety and Effectiveness of Abatacept in Psoriatic Arthritis Participants
Acronym: ALTEA
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-675
Record Dates: First submitted 2018-01-24; First posted 2018-02-01 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Psoriatic Arthritis (PsA)
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: naïve of abatacept, other biologic agents and Targeted synthetic disease modifying anti-rheumatic drugs (tsDMARDs)
- Cohort 2: "naïve of abatacept, who previously failed one tumor necrosis factor inhibitor (TNFi), but are naïve of any other biologic agent and tsDMARDs"
- Cohort 3: naïve of abatacept, who previously failed treatment with tsDMARDs and/or biologic agents** other than a single TNFi

SUMMARY:
The purpose of this study is a long-term, observational study of Abatacept in patients with Psoriatic Arthritis, a chronic inflammatory disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years or older
* Participants who signed an informed consent
* Participants diagnosed with PsA as per the criteria of the Classification of Psoriatic Arthritis (CASPAR) Study Group18
* Participants naïve of abatacept and who at their physician's discretion initiate abatacept
* Participants meeting criteria for abatacept treatment for PsA as specified in the German label

Exclusion Criteria:

* Participants who are currently included in any interventional clinical trial in PsA/Rheumatoid Arthritis (RA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population targeted by the study consists of patients with PsA that initiate treatment with abatacept
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Disease Activity index for PSoriatic Arthritis (DAPSA) | 12 months

SECONDARY OUTCOMES:
Participant retention rate | 12 Months
Proportion of concomitant treatment given | 12 Months
Initial dosage of Abatacept given | At Treatment Initiation
Frequency of Abatacept administration | 12 months
Descriptive Analysis: Reasons for Abatacept initiation | up to 2 years prior to treatment
Proportion of patients previously receiving by type of Disease modifying anti-rheumatic drug (DMARD) | up to 2 years prior to treatment
Descriptive Analysis: Socio-Demographics at Treatment Initiation | At Treatment Initiation
Descriptive Analysis: Disease history at Treatment initiation | Prior to treatment
Incidence of Risk factors and Comorbidities | At Treatment Initiation
Descriptive Analysis: Baseline Characteristics | up to 2 years prior to treatment
Descriptive Analysis: Change in participant characteristics and symptoms | 12 months
Proportion of Rheumatologist: Geography | up to 2 months prior to treatment to 12 months post treatment
Proportion of Rheumatologist: Type of Institution | up to 2 months prior to treatment to 12 months post treatment
Proportion and type of treatment after abatacept discontinuation | 12 months
Proportion of reasons for abatacept discontinuation and initiation of new therapy | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Nuremberg, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html